CLINICAL TRIAL: NCT03793322
Title: The Application of Indocyanine-Green(ICG) Fluorescence Imaging in Hepatocellular Carcinoma
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Zhujiang Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 201803
Record Dates: First submitted 2019-01-02; First posted 2019-01-04 (Actual); Last update posted 2019-01-04 (Actual); Status verified 2017-01

CONDITIONS: Hepatocellular Carcinoma
Keywords: Hepatocellular Carcinoma; Indocyanine-Green(ICG)
MeSH Terms: conditions — Carcinoma, Hepatocellular | interventions — Indocyanine Green

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Indocyanine-Green(ICG) injection group (Experimental)
  Interventions: Drug: Indocyanine-Green(ICG)

INTERVENTIONS:
Drug: Indocyanine-Green(ICG) — ICG was administered intravenously 24 hours before the operation , or directly into the portal vein branches supplying the tumor-bearing hepatic segment, after puncturing of the target segments under intraoperative ultrasonography guidance.

SUMMARY:
This study aims to evaluate the feasibility of indocyanine green (ICG)-based fluorescence imaging in the detection of liver tumors. By correlating the ICG fluorescence patterns with pathologically confirmed tumors , it would be possible to use fluorescence navigation system in helping promoting oncology treatment.

ELIGIBILITY:
Inclusion Criteria:

* 18 years≤ Age ≤70 years
* Compling with the diagnosis criteria of hepatic carcinoma.
* Primary hepatic carcinoma without intrahepatic or extrahepatic extensive cancer metastasis, the metastatic hepatic carcinoma whose primary focal has been controlled.
* Preoperative liver function is Child - Pugh grade A or B.
* The patients are volunteered for the study.

Exclusion Criteria:

* Patients with mental illness.
* Patients can't tolerate the operation owe to a variety of basic diseases (such as severe cardiopulmonary insufficiency, renal insufficiency, cachexia and blood system diseases, etc.
* The patients refused to take part in the study.
* There are other co-existed malignant tumors.
* Benign liver diseases.
* Indocyanine green allergy

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2017-01-01 (Actual); Primary Completion 2020-01-01 (Estimated); Study Completion 2020-12-31 (Estimated)

PRIMARY OUTCOMES:
The accuracy of detecting small liver tumor by ICG fluorescence. | 3 Days
  The tumor which aggregate ICG fluorescence will be resected and dignosed by pathology. The accuracy of detecting small liver tumor by ICG fluorescence will be evaluated.
The accuracy of positive margins of resection detected by ICG fluorescence. | 3 Days
  The surgery margins will be detected by ICG fluorescence. If there is fluorescence aggregating, we consider the presence of residual tumor in the margin and proven by histological examination.

CONTACTS AND LOCATIONS:
Overall Officials: Chihua Fang, Principal Investigator — China, Guangdong Zhujiang Hospital of The Southern Medical University
Locations (1):
- Zhujiang Hospital of Southern Medical University, Guangzhou, Guangdong, China